CLINICAL TRIAL: NCT02206789
Title: Evaluation of the Efficacy of 2% Cyclosporine in Preventing Graft Rejection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aravind Eye Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2011011CLI
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2011-10

CONDITIONS: Corneal Graft Rejection
MeSH Terms: interventions — prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- penetrating keratoplasty (Active Comparator): each arm will have two groups A and B.. Only on topical steroids(prednisolone acetate1%) group A On topical steroids + 2% cyclosporine Group B . Methodology of drug administration In both agroups 1. Schedule of topical steroid administration : 6 times for 2 weeks; 5 times for 2 weeks; 4 times for a month; 3 times for a month, and, subsequently twice-a-day until 1 year is completed . Topical steroids will be withdrawn at the end of ine year.Systemic steroids may be administered in the initial 2 weeks at the discretion of the investigators.
  3. Patients randomized to receive 2% cyclosporine will receive the same 3 times a day for 2years
  .
  Interventions: Drug: Prednisolone acetate1%,; Drug: Prednisolone acetate1%, cyclosporine 2%
- therapeutic keratoplasty (Active Comparator): each arm will have two groups A and B.. Only on topical steroids(prednisolone acetate1%) group A On topical steroids + 2% cyclosporine Group B . Methodology of drug administration In both agroups 1. Schedule of topical steroid administration : 6 times for 2 weeks; 5 times for 2 weeks; 4 times for a month; 3 times for a month, and, subsequently twice-a-day until 1 year is completed . Topical steroids will be withdrawn at the end of ine year.Systemic steroids may be administered in the initial 2 weeks at the discretion of the investigators. (For all patients with fungal keratitis topical steroids will be administered only after 2 weeks post keratoplasty.) Until then diclofenac sodium0.1% may be used 3. Patients randomized to receive 2% cyclosporine will receive the same 3 times a day for 2years
  .
  Interventions: Drug: Prednisolone acetate1%,; Drug: Prednisolone acetate1%, cyclosporine 2%

INTERVENTIONS:
Drug: Prednisolone acetate1%, — efficacy of prednisolone acetate1%alone versus prednisolone acetate 1%and cyclosporine 2% in preventing graft rejection
  Other Names: pred forte (Prednisolone acetate1% )
Drug: Prednisolone acetate1%, cyclosporine 2% — penetrating keratoplasty--efficacy of prednisolone acetate1%alone versus prednisolone acetate 1%and cyclosporine 2% in preventing graft rejection
  Other Names: pred forte (Prednisolone acetate1% ); aurosporine (cyclosporine 2%)

SUMMARY:
Aim/ Objective: Study consists of 2 separate and distinct entities A. Evaluation of the efficacy of 2% cyclosporine in preventing graft rejection in primary grafts w/o high risk characteristics study 1 (PKP study) B. Evaluation of the efficacy of 2% cyclosporine in preventing graft rejection in therapeutic keratoplasty- study 2(TKP study) Materials & Methods: In both arms Patients requiring keratoplasty, above the age of 18 whom satisfactorily meet The inclusion criteria are different for each study Eligible candidates will be enrolled after signing an Informed Consent form Patients will be randomized into one of 2 groups

* Only on topical steroids group A
* On topical steroids + 2% cyclosporine Group B Study design: Prospective, randomized non-blinded study at a single centre. Methodology In both arms

  1. Schedule of topical steroid administration : 6 times for 2 weeks; 5 times for 2 weeks; 4 times for a month; 3 times for a month, and, subsequently twice-a-day until 1 year is completed Systemic steroids may be administered in the initial 2 weeks at the discretion of the investigators. (For all patients with fungal keratitis topical steroids can preferrably be administered only after 2 weeks post keratoplasty.) Until then voveran ophtha may be used

  3. Patients randomized to receive 2% cyclosporine will receive the same 3 times a day for 2years

  4. All patients will be followed for a minimum period of 2 years

  5. Follow up schedule - at 1 week, 2 weeks, 1 month, 2 months, 3 months, then every 3 months until 2 years are completed

  6. All episodes of graft rejection will be treated as per accepted norms and the patient will no longer follow the standardized protocol for steroid administration

ELIGIBILITY:
Inclusion Criteria:

* FOR ARM 1

Age greater than 18 years

Vision more than 6/60 in the fellow eye.

No prior keratoplasty

Not more than 1 quadrant of corneal vascularisation

No peripheral anterior synechiae.

No active ocular surface disease (VKC, dry eye,)

Uncontrolled uveitis or glaucoma

No limbal stem cell failure.

No Prior h/o HSV

Primarily patients with dystrophies, degenerations and pseudophakic bullous keratopathy and non vascularised non herpetic corneal scars will be enrolled

ARM 2:

Inclusion criteria as above &

Those patients with medically unresponsive keratitis with no limbal involvement and in whom the graft size can be restricted to less than 9mm will be included in the study. This is to ensure that postoperative issues such as synechiae, recurrence of infection and uncontrolled glaucoma do not affect the study. Grafts must also be clear at the end of one month after surgery for patients to continue in the study..

Expected Outcome

1. Incidence of graft rejection in both arms.
2. secondary outcome Recovery from graft rejection in both arms.
3. Secondary outcomes- incidence of glaucoma and cataract.
4. secondary outcome Incidence of graft rejection in patients maintained only on cyclosporine after 1year.
5. It is expected that patients receiving cyclosporine will have a lesser incidence of graft rejection and exhibit faster recovery. The efficacy of long term prophylaxis of only cyclosporine in preventing graft rejection will also be evaluated.

Exclusion Criteria:Any condition that would increase the risk of non-rejection graft failure such as Stevens-Johnson syndrome, xerophthalmia or severe exposure keratitis. Schirmer's test ≤ 5 mm in 1 minute Clinical evidence of limbal stem cell deficiency History of or active herpes simplex virus keratitis or other acute corneal infection

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
graft rejection | 5 years

SECONDARY OUTCOMES:
recovery from graft rejection | 5 years
Incidence of graft rejection in patients maintained only on cyclosporine after 1year | 5 years
  .graft rejection in patients only on cyclosporine 2% eye drops in the second year of study

OTHER OUTCOMES:
incidence of glaucoma and cataract. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Anita Raghavan, Principal Investigator — Medical Cornea Consultant
Locations (1):
- Dr.Anita Raghavan, Coimbatore, Tamil Nadu, India